CLINICAL TRIAL: NCT05497947
Title: Evaluation of the French Translation of Swallowing (SOAL-VF) Patient Reported Outcomes (PRO) After Total PharyngoLaryngectomy
Acronym: SOAL-VF
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Valence (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH-CHV-05
Record Dates: First submitted 2022-08-10; First posted 2022-08-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pharyngeal Cancer; Swallowing Disorder; Larynx Cancer
Keywords: SOAL; patient reported outcomes
MeSH Terms: conditions — Pharyngeal Neoplasms; Deglutition Disorders; Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A monocentric study to evaluate the french translation of Swallowing (SOAL-VF) Patient Reported Outcomes (PRO) after Total PharyngoLaryngectomy

DETAILED DESCRIPTION:
the SOAL questionnaire is a validated Patient Reported Outcomes (PRO) questionnaire in English language.

The aim of this study is to develop a new tool in french language and to evaluate incidence and the specific impact of swallowing disorders on the quality of life of patients after Total PharyngoLaryngectomy.

ELIGIBILITY:
Inclusion Criteria:

* Total PharyngoLaryngectomy
* Age ≥ 18 years old
* Read, write and understand the French language

Exclusion Criteria:

* Patient under guardianship, deprived of liberty, safeguard of justice
* Refusal to participate in research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated by Total PharyngoLaryngectomy in CH Valence
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
SOAL- VF | up to 6 months
  Patient reported outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BUIRET, MD, Principal Investigator — CH VALENCE
Locations (1):
- Ch Valence, Valence, Drome, France

IPD SHARING:
Plan to Share IPD: Undecided